CLINICAL TRIAL: NCT06989957
Title: Psilocybin and MDMA for Post-traumatic Stress Disorder (PTSD)
Brief Title: Psilocybin and Methylenedioxymethamphetamine (MDMA) for Post-traumatic Stress Disorder (PTSD)
Acronym: PAM-VET
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Gracias Family Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00463389
Record Dates: First submitted 2025-05-12; First posted 2025-05-25 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Posttraumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Psilocybin; N-Methyl-3,4-methylenedioxyamphetamine

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, active control study comparing a single dose of co-administered MDMA + psilocybin (exact dosages not disclosed) with a single dose of co-administered MDMA active placebo + psilocybin active placebo (exact dosages not disclosed)
Who Masked: Participant, Investigator
Masking Description: The first dosing session will be double-blind; the second dosing session will be single-blind (participant masked).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Experimental MDMA + psilocybin (exact dosage not disclosed) (Experimental): MDMA will be given initially, followed by psilocybin 30 minutes later.
  Interventions: Drug: Psilocybin; Drug: MDMA
- Comparator MDMA + psilocybin (exact dosage not disclosed) (Active Comparator): MDMA will be given initially, followed by psilocybin 30 minutes later.
  Interventions: Drug: Psilocybin; Drug: MDMA

INTERVENTIONS:
Drug: Psilocybin — Experimental Psilocybin (exact dosages not disclosed)
  Arms: Experimental MDMA + psilocybin (exact dosage not disclosed)
Drug: Psilocybin — Comparator Psilocybin (exact dosages not disclosed)
  Arms: Comparator MDMA + psilocybin (exact dosage not disclosed)
Drug: MDMA — Experimental MDMA (exact dosages not disclosed)
  Arms: Experimental MDMA + psilocybin (exact dosage not disclosed)
Drug: MDMA — Comparator MDMA (exact dosages not disclosed)
  Arms: Comparator MDMA + psilocybin (exact dosage not disclosed)

SUMMARY:
The purpose of this study is to assess the safety and effectiveness of co-administered MDMA and psilocybin in military Veterans with a diagnosis of Posttraumatic Stress Disorder (PTSD).

To apply or learn more, please view our website: https://hopkinspsychedelic.org/pamvet

DETAILED DESCRIPTION:
The proposed randomized, double-blind, active control study will compare a single experimental dose of co-administered MDMA + psilocybin (exact dosages not disclosed) with a single comparator dose of co-administered MDMA + psilocybin (exact dosages not disclosed). For the co-administered dosing session, MDMA will be given initially, followed by psilocybin 30 minutes later. Approximately 1.5 months after the first dosing session, a second single-blind (participant masked) dosing session will occur. The study will recruit adult Veterans with PTSD for ≥ 6 months.

ELIGIBILITY:
Inclusion Criteria:

* >=21 years old
* Military Veteran
* Have given written informed consent
* Able to swallow pills
* Have a confirmed DSM-5 diagnosis of Post-traumatic Stress Disorder with symptom duration >= 6 months
* Have a baseline CAPS-5 score of >=28
* Be judged by study team clinicians to be at low acute risk for suicidality
* Concurrent psychotherapy is allowed if the type and frequency of the therapy has been stable for at least two months prior to screening and is expected to remain stable during participation in the study.
* Be medically stable as determined by screening for medical problems via a personal interview, a medical questionnaire, a physical examination, an electrocardiogram (ECG), and routine medical blood and urinalysis laboratory tests
* Agree to consume approximately the same amount of caffeine-containing beverage (e.g., coffee, tea) that he/she consumes on a usual morning, before arriving at the research unit on the mornings of drug session days. If the participant does not routinely consume caffeinated beverages, he/she must agree not to do so on session days.
* Agree to refrain from using any psychoactive drugs, including alcoholic beverages within 24 hours of each drug administration. The exceptions are caffeine and nicotine.
* Agree to refrain from using any caffeine or nicotine within 2 hours of dosing session start.
* Agree not to take any as needed (PRN) medications on the mornings of drug sessions without approval of the treatment team.
* Agree not to take sildenafil (Viagra®), tadalafil, or similar medications within 72 hours of each drug administration.
* Agree to stop taking 5HT2A antagonist medications at least 5 half-lives before dosing.
* Agree that for one week before each drug session, he/she will refrain from taking any nonprescription medication, nutritional supplement, or herbal supplement except when approved by the study investigators. Exceptions will be evaluated by the study investigators and will include acetaminophen, non-steroidal anti-inflammatory drugs, and common doses of vitamins and minerals.
* Have no lifetime use of serotonin 2A receptor (5-HT2A) agonist hallucinogens and/or MDMA at a greater dosage than a level typically defined as 'microdose.'
* Have at least a high school level of education or equivalent (e.g. GED).
* Weigh between 40kg- 120kg.
* Must provide a contact (relative, spouse, close friend or other support person) who is willing and able to be reached by the investigators in the event of a participant becoming suicidal or unreachable
* Agree to be released into the custody of a close friend or family member who has agreed to take charge of the study participant as a condition of leaving the testing facility, or agree to be accompanied home or to an accommodation by a member of the study team
* May have a history of or current Diabetes Mellitus (Type 2) if additional screening measures rule out underlying cardiovascular disease, if the condition is judged to be stable on effective management, and with approval by the Medical Monitor
* May have hypothyroidism if taking adequate and stable thyroid replacement medication
* May have a history of, or current, glaucoma if approval for study participation is received from an ophthalmologist

Exclusion Criteria:

* Current or past history of meeting DSM-5 criteria for schizophrenia spectrum or other psychotic disorders (except substance/medication-induced or due to another medical condition), or Bipolar I or II Disorder
* Current or history within one year of meeting DSM-5 criteria for a moderate or severe alcohol, or other drug use disorder (excluding tobacco, caffeine, and cannabis)
* Current or history within one year of meeting DSM-5 criteria for Borderline Personality Disorder.
* Clinically significant suicidal ideation (e.g. with strong intent or means; C-SSRS > 3) within past 6 months
* Have a first degree relative with schizophrenia or other psychotic disorders (except substance/medication-induced or due to another medical condition), or bipolar I disorder
* Nicotine dependence that would be incompatible with an individual to be nicotine free for 8-10 hours on a dosing session day
* Medical condition incompatible with MDMA or psilocybin administration (e.g., cardiovascular, drug-induced hyperthermia, hyponatremia).
* Currently taking on a daily basis any medications (including herbal substances and supplements) with a Central Nervous System effect on serotonin (including serotonin-reuptake inhibitors (SRIs), monoamine oxidase inhibitors (MAOIs)), or any medications that affect liver enzyme (2D6) metabolism (e.g., Bupropion)
* Currently taking efavirenz, Acetaldehyde dehydrogenase inhibitors such as disulfiram (Antabuse), Alcohol dehydrogenase inhibitors, uridine diphosphate glucuronosyltransferase enzyme (UGT1A9) inhibitors or UGT1A10 inhibitors such as phenytoin, regorafenib, eltrombopag.
* On unstable/changing dose of opioid, benzodiazepine or other psychoactive or pain medication within 4 weeks prior to enrollment and/or unable to abstain from medication on drug administration day
* Current use/positive toxicology for illicit drugs; or positive breath alcohol test at screening and/or prior to each drug administration session
* Lifetime use of any psychedelic drug (e.g., MDMA, psilocybin) at a dosage greater than a level typically defined as 'microdose.'
* Clinically significant transaminitis (aspartate aminotransferase (AST) or alanine aminotransferase (ALT) greater than two times normal value).
* Women who are pregnant (as indicated by a positive urine pregnancy test assessed at intake and before each drug session) or nursing;
* Women who are of child-bearing potential and sexually active agree to use highly effective means of birth control (i.e. implants, injectables, combined oral contraceptives, progestin-containing intrauterine device (IUD) or vasectomised partner) for the duration of this study.
* Cardiovascular conditions: coronary artery disease, stroke, angina, uncontrolled hypertension, a clinically significant ECG abnormality (e.g., atrial fibrillation), prolonged corrected QT interval (QTc) (i.e., QTc > 450 msec), heart valve, or transient ischemic attack (TIA) in the past year.
* History of seizures and/or epilepsy with history of seizures.
* Type 1 diabetes.
* BMI < 18
* Are likely, in the investigator's opinion and via observation during the Preparatory Period, to be re-exposed to the index trauma or other significant trauma in daily life, lack social support, or lack a stable living situation.
* Have received Electroconvulsive Therapy (ECT) within 12 weeks of enrollment
* Have a history of any medical condition that could make receiving a sympathomimetic drug harmful because of increases in blood pressure and heart rate. This includes, but is not limited to, a history of myocardial infarction, cerebrovascular accident, or aneurysm.

  * Participants with other mild, stable chronic medical problems may be enrolled if the site physician and investigators agree the condition would not significantly increase the risk of MDMA administration or be likely to produce significant symptoms during the study that could interfere with study participation or be confused with side effects of the study drugs. Examples of stable medical conditions that could be allowed include, but are not limited to Diabetes Mellitus (Type 2), Human Immunodeficiency Virus (HIV) infection, Gastroesophageal Reflux Disease (GERD), etc.
* Any medical disorder judged by the investigator to significantly increase the risk of MDMA administration by any mechanism would require exclusion
* Have symptomatic liver disease or significant liver enzyme elevations

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09-17 (Actual); Primary Completion 2028-08 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events | 30 weeks
  Participants will be asked how the participant has been feeling since the last visit and will be asked about incidence of any adverse events (AEs) since the last visit. In addition to monitoring any spontaneously reported AEs at each study visit, participants will also be queried specifically if the participant has experienced any return of drug-like (i.e., MDMA or psilocybin) effects or other AEs the participant suspects to be drug-related at all meetings occurring after the first dosing session. A serious adverse event (SAE) will be defined as either: a death or a life-threatening occurrence, including hospitalization; incarceration; new onset of a significant medical disorder; or significant exacerbation of an existing medical disorder. All AEs and SAEs will be monitored closely by the study team to guide appropriate follow-up and all AEs and SAEs will be documented and followed to resolution.
The Columbia Suicide Severity Rating Scale (C-SSRS) | 33 weeks
  The Columbia Suicide Severity Rating Scale (C-SSRS) will be used to assess severity of suicide ideation during every study visit. Suicidal Ideation Intensity scale (0-25 score range summed from five items, with higher scores indicating more severe suicidal ideation).
Clinician-Administered PTSD Scale for Diagnostic and Statistical Manual-5 (CAPS-5) | 33 weeks
  The CAPS-5 assessment consists of 30 items that are designed to measure the frequency and intensity of PTSD symptoms, covering all 20 Diagnostic and Statistical Manual-5 (DSM-5) PTSD symptoms. Each item is scored on a 5-point scale (0, absent - 4, extreme/incapacitating). Score ranges from 0 to 80 with higher scores indicating higher symptom severity.
PTSD Checklist (PCL-5) | 33 weeks
  The PTSD Checklist for DSM-5 is a self-report psychometric instrument widely employed in both clinical and research settings to assess the presence and severity of PTSD symptoms as outlined in the DSM-5. The PCL-5's 20 items correspond to the DSM-5 symptom criteria for PTSD. This version of the PCL-5 will assess symptoms within the preceding week. PCL-5 questionnaires will be administered to participants via email (not clinician-administered). It is scored by summing the responses to 20 items, each rated on a 5-point scale (0-4), resulting in a total score ranging from 0 to 80. A higher score indicates greater severity of PTSD symptoms.
World Health Organization Quality of Life- Brief version (WHOQOL-BREF) | 33 weeks
  The World Health Organization Quality of Life (WHOQOL) Brief version scores on this subscales range from 0-30 with higher scores reflecting better quality of life.

SECONDARY OUTCOMES:
Clinical Global Impression (CGI-I) Scale | 9 weeks
  The CGI-I scale ranges from 1 to 7 (1=very much improved; 2=much improved, 3=minimally Improved, 4=no change, 5=minimally worse, 6= much worse, and 7=very much worse).
Patient global impression of improvement (PGI-I) | 9 weeks
  The PGI-I was developed for use in National Institute of Mental Health sponsored clinical trials in order to broadly define participant progress/improvement. The PGI-I scale is a 7-point scale used to assess a patient's perception of condition's change, typically after a treatment or intervention. The scale ranges from 1 to 7, with 1 representing "very much improved" and 7 representing "very much worse."
The Sheehan Disability (SDS) Scale | 33 weeks
  The Sheehan Disability (SDS) Scale will be used to assess functional impairment in three domains of disability that can be impaired during depression: work/school, social, and family life. It uses a Likert scale from 0 to 10, with higher scores indicating greater functional impairment. The total SDS score ranges from 0 to 30.

CONTACTS AND LOCATIONS:
Overall Officials: Brandon Weiss, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Center for Psychedelic and Consciousness Research, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No